CLINICAL TRIAL: NCT04139512
Title: One-abutment One-time for Immediate Restoration Procedure in the Esthetic Zone: A Randomized Controlled Trial Comparing Conventional Versus Full Digital Workflow
Brief Title: One-abutment One-time for Immediate Restoration Procedure in the Esthetic Zone
Acronym: IONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Professor , doctor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B707201731117
Record Dates: First submitted 2019-08-19; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Implant Tissue Failure
MeSH Terms: interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Intervention Model Description: The present study was designed as a randomized controlled trial comparing immediate restoration procedure in the esthetic zone with a one abutment one-time technique and using a conventional (control group) versus full digital workflow (test group),
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- guided surgery (Other): test group, using a full digital workflow procedure
  Interventions: Procedure: guided surgery
- conventional technic (Other): free- hand technic to place implant
  Interventions: Procedure: conventionnel implant placement

INTERVENTIONS:
Procedure: guided surgery — placement of implant with local anesthesia using full guided surgery protocol versus free- hande one
  Arms: guided surgery
Procedure: conventionnel implant placement — placement of dental implant with conventionnal freehand technic
  Arms: conventional technic

SUMMARY:
Objectives: The aim of this randomized control trial was to compare immediate restoration procedure with a one abutment one-time technique using a conventional versus full digital workflow. Surgical accuracy, provisional fit and patient reported outcome measures (PROMs) of.

DETAILED DESCRIPTION:
Objectives: The aim of this randomized control trial was to compare immediate restoration procedure with a one abutment one-time technique using a conventional versus full digital workflow. Surgical accuracy, provisional fit and patient reported outcome measures (PROMs) of.

Material and method: Sites with single edentulous spaces and neighboring natural teeth were randomized into static computer-aided implant surgery (s-CAIS) or freehand placement implant surgery groups. In both groups, digital implant planning was performed using data from cone beam computed tomography (CBCT) and surfaces scans. In the s-CAIS group, a surgical guide was produced and used for fully guided implant surgery, while in the freehand group, the implants were placed in a freehand manner. the deviations in angles, shoulders and apexes between planned and actual implant positions were measured based on postoperative optic impressions. In the test group, a custom-made zirconia abutment and a provisional restoration were immediately placed using a full digital workflow whereas in the control group, a physical impression was taken, and the abutment and crown were placed 10 days post-surgery. Loading outcomes (interproximal contact, occlusal contact, white esthetic score (WES)) were assessed as the PROMs.

ELIGIBILITY:
Inclusion criteria

* Subjects must have voluntarily signed the informed consent form before any study related action
* Age > 18 years old
* Single missing tooth or 2 non-adjacent missing teeth in the aesthetic area of the upper jaw. Patients who require an extraction and immediate implant placement can be included.
* Men/women
* Good systemic health (ASA I/II)
* No contra indication against oral surgical interventions
* At least 10 mm in the vertical dimension
* At least 7 mm in the bucco-palatal dimension
* No need for simultaneous bone augmentation procedure. However, a bone augmentation could have been realized 4 months prior to the digital planning of the surgery
* Healthy periodontal condition and full mouth plaque score (FMPS) lower or equal than 25%

Exclusion criteria

* Autoimmune disease requiring medical treatment
* Medical conditions requiring prolonged use of steroids
* Use of bisphosphonates intravenously or more than 3 years of oral use
* Infection (local or systemic) Each infection will be evaluated prior to study procedure for suitability. Patients with gingivitis or local infection will undergo a medical treatment prior to its entrance to the study.

In case of systemic infection, the evaluation will be based on medical anamneses and, if necessary, will be referred to relevant medical tests.

* Current pregnancy or breastfeeding women
* Alcoholism or chronically drug abuse
* Immunocompromised patients
* Uncontrolled diabetes
* Smokers, more than 10 cigarettes per day

Local exclusion criteria

* Untreated local inflammation
* Mucosal disease or oral lesions
* History of local irradiation therapy in the head-neck area
* Persistent intraoral infection
* Patients with bad oral hygiene or unmotivated for normal home care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the surgical accuracy | The day of the surgery
  The STL files (stereolithography files) were superimposed with pre-operative CBCT (Cone beam computed tomography) images using automated surface best fit matching with the iterative closest point algorithm in the treatment evaluation mode, coDiagnostiX® software version 9.7 (Dental Wings Inc). The mean deviations at the implant shoulder and apex between the planned and actual implant positions were measured in millimeters (mm), as well as the divergence of the implant axis in degrees. All measurements were performed by a single dentist, who conducted the virtual implant planning in all cases.
Clinical fit of the provisional restoration measurements | 10 days post surgery
  The measurements were based on the adaptation of the provisional crown. Interproximal contacts were evaluated according to the criteria described by Syrek (Syrek et al., 2010). Dental floss (Johnson & Johnson Reach®, Waxed dentotape, New Brunswick, NJ, USA) was used to check the interproximal contact. A score from 1 to 4 was given to the fitting criteria (the higher the score, the better the adaptation).

SECONDARY OUTCOMES:
WES | 10 days post surgery
  To evaluate the esthetic outcomes of the provisional crown, the White Esthetic Score (WES) was reported. The highest WES score was 10, which represented a close match with the clinical single-tooth crown present at the contralateral natural tooth or neighboring teeth. The WES was evaluated by a blinded prosthodontic, based on photography.
Patient-reported outcomes measures (PROMs) | 10 days post surgery
  PROMs were obtained using a VAS form immediately after the immediate restoration of the implant. Five questions were used:
  1. Do you feel your provisional tooth as a natural tooth? (0 = not at all to 10, absolutely).
  2. Do you find your provisional tooth looks like a natural tooth? (0 = not at all to 10, absolutely).
  3. How much discomfort did you feel during the physical impression? (0 = little or 10, a lot) for the control group.
     How much discomfort did you feel during the optical impression? (0 = little to 10, a lot) for the test group.
  4. Would you be willing to undergo this treatment again? (0= not at all to 10, absolutely).
  5. Are you satisfied with the aesthetics outcomes of your provisional tooth. (0 = not at all to 10, absolutely).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège - Service de Médecine Dentaire, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No